CLINICAL TRIAL: NCT01208012
Title: Impact of Liraglutide on Endothelial Function and Microvascular Blood Flow in Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ikfe-CRO GmbH (Industry)
Collaborators: Novo Nordisk A/S (Industry); IKFE Institute for Clinical Research and Development (Other)
Responsible Party: Prof. Thomas Forst, MD, ikfe GmbH
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Lira-Vasc-001
Record Dates: First submitted 2010-09-17; First posted 2010-09-23 (Estimated); Last update posted 2011-03-15 (Estimated); Status verified 2011-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus treatment Metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (No Intervention): Patients taking Metformin at individual dose
- Metformin and Liraglutide (Experimental): Patients taking Metformin at individual dose and Liraglutide 0.6 mg once daily for the 1st week, 1.2 mg daily for another 5 weeks, 1.8 mg daily for another 6 weeks.
  Interventions: Drug: Victoza®

INTERVENTIONS:
Drug: Victoza® — Patients taking Metformin at individual dose and Liraglutide 0.6 mg once daily for the 1st week, 1.2 mg daily for another 5 weeks, 1.8 mg daily for another 6 weeks. When arrived at the dosage of 1.8 mg daily and the dose is not tolerated by the patient, the dose of Liraglutide can be decreased.Liraglutide is injected in the subcutaneous tissue once daily
  Other Names: Victoza®, Liraglutide
  Arms: Metformin and Liraglutide

SUMMARY:
The trial is a phase IV clinical trial investigating the impact of Liraglutide on endothelial function and microvascular blood flow in 44 patients with type 2 diabetes mellitus aged 30-65 and HbA1c ranging from ≥ 5.5% ≤ 7.0%. The patients will be randomized into two study arms, one arm will be treated with Metformin monotherapy, the second arm will be treated with Metformin and Liraglutide at an increasing dose (0.6 mg/day to 1.8 mg/day.)

DETAILED DESCRIPTION:
Type 2 Diabetes Mellitus (DM) is associated with increased cardiovascular risk and the majority of type 2 diabetic patients die due to the vascular complications of Diabetes Mellitus. In type 2 diabetic patients, an early marker in the biogenesis of atherosclerosis and cardiovascular disease is the occurrence of endothelial dysfunction with subsequent deterioration in micro- and macrovascular blood flow and tissue supply. Also several mechanistic pathways linking Diabetes Mellitus with endothelial dysfunction and cardiovascular complications are postulated. Recent studies aimed to investigate the vasoprotective effect of strict glycaemic control using conventional treatment algorithms failed to reduce cardiovascular risk in patients with Diabetes Mellitus type 2. Numerous pharmacological drugs are available to reduce blood glucose levels in type 2 diabetic patients. Beside comparable glucose lowering efficacy, some of them evolve limited or even adverse effects on vascular function and cardiovascular risk. Therefore, ideally new treatments in Diabetes Mellitus type 2 provide more than just reducing blood glucose values. Future treatments in type 2 Diabetes Mellitus will be judged on their potency to affect the cardiovascular risk profile in patients with Diabetes Mellitus type 2.

Liraglutide is a Glucagon-like peptide-1 (GLP-1) analogue shown to be effective in the treatment of type 2 Diabetes Mellitus. Liraglutide was shown to improve blood glucose levels not only by stimulating insulin secretion from the β cell, but also by improving the conversion of intact proinsulin into insulin and C-peptide in the granula of the β cell. While in rodents, GLP-1 and its analogues showed an increase in β cell regeneration and an inhibitory effect on β cell apoptosis, the effect of GLP-1 analogues on β cell mass in humans is less clear. Beyond its effects on β cells, Liraglutide and other GLP1 analogues were shown to suppress the glucagon release from α cells and to evolve a supportive effect on weight reduction by central and probably peripheral effects.

Beside these effects of GLP-1-analogues on β cell physiology and glucose metabolism, recent studies suggested several pleiotrophic effects of GLP-1 treatment which go beyond glycaemic control. Receptors for GLP-1 have been located in myocardial and endothelial cells, and GLP-1 supplementation was found to improve myocardial and endothelial function in diabetic and in non-diabetic subjects. In endothelial cells, isolated from human coronary arteries, GLP-1 rapidly activates endothelial nitric oxide synthase (eNOS) and stimulates nitric oxide (NO) production, promotes cell proliferation and inhibits glucolipoapoptosis. In addition, in transformed vascular endothelial cells, GLP-1 protects endothelial dysfunction incurred by tumor necrosis factor-α (TNF-α) through the modulation of the expression of vascular adhesion molecules and plasminogen activator inhibitor-1 (PAI-1). Chronic administration of GLP-1 analogues is associated with a significant reduction in blood pressure. Therefore it seems conceivable, that in patients with Diabetes Mellitus type 2, treatment with the GLP-1 analog Liraglutide might improve the cardiovascular risk profile beyond glucose control by stimulating endothelial NO release and by improving endothelial function.

The goal of our study is to investigate the vascular and endothelial effects of adding Liraglutide treatment to type 2 diabetic patients previously treated with Metformin.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes Mellitus type 2
2. HbA1c ≥ 5.5% and ≤ 7.0%
3. Treatment with Metformin (daily dose 500 - 3000 mg monotherapy, the past 3 months)
4. Age 30 - 65 years

Exclusion Criteria:

1. Pre-treatment with PPAR gamma agonists or DPP IV inhibitors or GLP-1 analogues within the last three months
2. History of type 1 Diabetes Mellitus
3. No full legal mental and physical ability to give informed consent
4. Uncontrolled hypertension (systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 90 mmHg)
5. Anamnestic acute and chronic infections
6. Inflammatory bowel disease and/or diabetic gastroparesis
7. Anamnestic history of epilepsy
8. Anamnestic history of hypersensitivity to the study drugs or to drugs with similar chemical structures
9. History of severe or multiple allergies
10. Treatment with any other investigational drug within 3 months before trial entry
11. Progressive fatal disease
12. History of drug or alcohol abuse in the past 2 years
13. Liver disease with ASAT or ALAT above 3 times the upper normal limit
14. Serum potassium > 5.5 mmol/L
15. Moderate to Severe Kidney disease with a GFR ≤ 60 ml/min
16. Pregnancy or breast feeding
17. Sexually active woman of childbearing potential not practicing a highly effective method of birth control as defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, hormonal IUDs, sexual abstinence or vasectomised partner
18. Have had more than one unexplained episode of severe hypoglycaemia (defined as requiring assistance of another person due to disabling hypoglycaemia) within 6 months prior to screening visit
19. History of dehydration, diabetic precoma, diabetic ketoacidosis or diabetic gastroparesis
20. Acute (within the previous 2 days) or scheduled investigation with iodine containing radiopaque material
21. Acute myocardial infarction, open heart surgery or cerebral event (stroke/TIA) within the previous 6 months
22. Anamnestic uncontrolled unstable angina pectoris, pericarditis, myocarditis, endocarditis, haemodynamic relevant aortic stenosis, aortic aneurysma or heart insufficiency NYHA III or IV
23. Anamnestic recent pulmonary embolism or pulmonary insufficiency
24. Smoking within the last 6 months (> 1 cigarette/day)
25. Planned change in antidiabetic, lipid lowering or blood pressure medication

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
The difference in increase of retinal blood flow after flicker stimulation of retinal endothelial cells | timepoint 0 and after 6 and 12 weeks
  Retinal capillary blood flow will be assessed using scanner laser doppler flowmetry.

SECONDARY OUTCOMES:
Central vascular elasticity | timepoint 0 and after 6 and 12 weeks
  Central arterial elasticity will be measured by Pulse wave velocity.
Skin endothelial function and Skin oxygenation | timepoint 0 and after 6 and 12 weeks
  Microvascular skin blood flow and postcapillary tissue oxygenation (sO2)will be measured.
Blood glucose control | timepoint 0 and after 6 and 12 weeks
  Fasting plasma glucose will be measured.
Blood glucose control | up to 2 weeks before baseline and after 6 and 12 weeks after baseline
  HbA1c will be maesured.
Change of biomarkers of sub-clinical inflammation and cardiovascular risk | timepoint 0 and after 6 and 12 weeks
  Biomarkers PAI-1, hsCRP, VCAM, E-selectin and ADMA will be measured.
Change of biomarker of heart failure | timepoint 0 and after 6 and 12 weeks
  NT-pro BNP will be measured.
Insulin/ intact Proinsulin ratio, C-peptide | timepoint 0 and after 6 and 12 weeks
  Insulin Intact Proinsulin and C-peptide will be maesured.
Change of body weight | up to 2 weeks before baseline and after 6 and 12 weeks after baseline
  Body weight will be measured.
Safety evaluation | up to 2 weeks before baseline and after 12 weeks post baseline
  The safety evaluation includes:
  * Metabolic parameters indicating hepatic function (ALAT, ASAT, γ-GT)
  * Blood analysis (Alkaline Phosphatase, Blood cell count)
  * Change in pancreas function (Amylase, Lipase)
  * Change in renal function (Creatinine, Potassium)
  * Change in thyroid function (Calcitonin)
  * Vital signs (Blood Pressure, Radial Pulse, ECG)
  * β-HCG (only female patients of childbearing potential)
  * Adverse Events
  * Adverse Drug Reactions

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Forst, Prof. Dr., Principal Investigator — Ikfe GmbH
Locations (1):
- IKFE Institute for Clinical Research and Development, Mainz, Germany

REFERENCES:
- [Derived] Forst T, Michelson G, Ratter F, Weber MM, Anders S, Mitry M, Wilhelm B, Pfutzner A. Addition of liraglutide in patients with Type 2 diabetes well controlled on metformin monotherapy improves several markers of vascular function. Diabet Med. 2012 Sep;29(9):1115-8. doi: 10.1111/j.1464-5491.2012.03589.x. PMID 22288732